CLINICAL TRIAL: NCT05897905
Title: A Feasibility Study Investigating an Early, Personalised, Follow-up Programme for People After Minor Stroke
Brief Title: Improving Follow up Care for People After Minor Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23CX8211
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Stroke, Acute
Keywords: Secondary prevention; Adjustment to life after stroke; Hidden impairments; Cognition; Mood; Fatigue
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): All participants will receive a brief routine stroke medical follow-up appointment.
- Personalised, holistic based follow-up appointments underpinned by self determination theory. (Experimental): Participants will receive two follow-up appointments at two and six weeks after discharge.
  Interventions: Behavioral: Personalised, holistic follow-up appointments underpinned by self determination theory

INTERVENTIONS:
Behavioral: Personalised, holistic follow-up appointments underpinned by self determination theory — Appointment 1 (two weeks after discharge):
  * Address participants knowledge gaps as regards their stroke, medication and secondary prevention.
  * Detailed biopsychosocial review.
  * Understand participant priorities and jointly set goals.
  * Agreeing onward referrals if needed.
  * Written summary sent to GP with copy to participant.
  Appointment 2 (six weeks):
  * Review priorities identified in post stroke review checklist.
  * Review goals and plans from first appointment.
  * Address any new or persistent information gaps.
  * Review hidden impairments that may be impacting on return to work, activities of daily living, relationships or general well-being.
  * Agreeing onward referrals and action plan.
  * Written summary and plan sent to GP.
  Arms: Personalised, holistic based follow-up appointments underpinned by self determination theory.

SUMMARY:
The goal of this feasibility study is to ascertain if this follow-up programme of care can feasibly be implemented within a healthcare system with people after minor stroke.

The main feasibility questions are:

i) To establish recruitment uptake ii) To establish treatment adherence iii) To determine participant retention. Participants will be randomly allocated to the intervention and control group. Those in the intervention group will receive a follow-up telephone call at two weeks after discharge and a second follow-up appointment at six weeks after discharge. Outcome measures will be taken at twelve weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18
* Clinical or radiological diagnosis of minor stroke from a stroke consultant.
* Admitted to HASU or seen in rapid assessment/TIA clinic.
* Pre-admission mRS of 0-3 with no formal package of care prior to stroke.
* Discharge mRS of 0-3.
* No onward referral to community therapy team or for package of care.
* Has capacity to consent.

Exclusion Criteria:

* Any serious co-morbidities that would impact a person's ability to participate in the follow-up appointments and outcome measurement.
* Insufficient English to engage in intervention and outcome measures and no family or friends to support with this.
* Not resident in England.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Proportion of participants randomised relative to the total number meeting the inclusion criteria.
Treatment completion rate | 6 weeks post randomisation
  Proportion of participants who attend both follow-up appointments
Retention rate | 12 weeks post randomisation
  Proportion of participants that complete the follow-up questionnaires

SECONDARY OUTCOMES:
PROMIS10 | 2 weeks and 12 weeks
  Patient reported outcome measures information system
Health Care Climate Questionnaire Short Form | Baseline and 12 weeks
  Patient reported outcome measure
MOCA | Baseline and 12 weeks
  Cognitive assessment
PHQ9 | 12 weeks
  Mood score
GAD7 | 12 weeks
  Anxiety score

OTHER OUTCOMES:
Qualitative interviews | 13 weeks
  Semi-structured

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crow, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No